CLINICAL TRIAL: NCT00322582
Title: Open Labeled of the Study the Genetic Basis for Familial Cardiomyopathy in Patients With Idiopathic
Brief Title: The Genetic Basis for Familial Cardiomyopathy in Patients With Idiopathic Cardiomyopathy
Status: Terminated | Type: Observational
Why Stopped: no financial resources were available to complete the study
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Offer Amir, Offer Amir, MD, Carmel Medical Center, Carmel Medical Center
Other Study IDs: GEN/ICM; 136-2005
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2007-01

CONDITIONS: Cardiomyopathy
Keywords: familial cardiomyopathy; genetics analysis
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples

SUMMARY:
In many of the patients with cardiomyopathy, the etiology is not clear . In about 30% there is a family history of cardiomyopathy .Our aim is to study the genetics basis for these patients with cardiomyopathy with no clear etiology and who have a first degree family relative with cardiomyopathy as well.

DETAILED DESCRIPTION:
A total of 950 blood samples will be collected from patients with idiopathic cardiomyopathy and their relatives and will be analysed for genetics analysis.

ELIGIBILITY:
Inclusion Criteria:

* history of cardiomyopathy
* etiology not known
* family history of cardiomyopathy
* ability to understand and sign the informed consent

Exclusion Criteria:

* refusal to participate
* pregnancy
* current participation in another active treatment study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: History of cardiomyopathy
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2007-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Offer Amir, MD, Study Director — Lady Davis Carmel Hospital
Locations (1):
- Carmel Medical Center, Haifa, Israel

REFERENCES:
- [Background] Murphy RT, Starling RC. Genetics and cardiomyopathy: where are we now? Cleve Clin J Med. 2005 Jun;72(6):465-6, 469-70, 472-3 passim. doi: 10.3949/ccjm.72.6.465. PMID 16018289